CLINICAL TRIAL: NCT06878105
Title: Evaluation of Fixed and Personal Assets for Patient Blood Management Implementation in CEE Countries in Practice
Brief Title: Patient Blood Management Implementation in CEE Study
Acronym: CEEPBM
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Dr. Fazakas János, Associate Professor, Semmelweis University
Other Study IDs: CG90142103
Record Dates: First submitted 2024-08-02; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Anemia; Coagulopathy
MeSH Terms: conditions — Anemia; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hospital self audit data baseline before PBM training: Anticipated 50 hospitals from Hungary, Romania, Czech Republic, Slovakia, Croatia, Austria. Only data about drugs/blood products used as medical routine will be recorded - no evaluation of any drug effect/efficacy.
  Interventions: Other: Data collection on interventions performs as per medical routine
- Hospital self audit data after 6 month after PBM training: Anticipated 50 hospitals from Hungary, Romania, Czech Republic, Slovakia, Croatia, Austria.Only data about drugs/blood products used as medical routine will be recorded - no evaluation of any drug effect/efficacy.
  Interventions: Other: Data collection on interventions performs as per medical routine

INTERVENTIONS:
Other: Data collection on interventions performs as per medical routine — No intervention other than routine medical practice

SUMMARY:
The goal of the study is data collection on available fixed and personal assets required for Patient Blood Management (elements of the 3 pillars of PBM) in Central Eastern Europe countries hospitals, status before and after PBM training.

DETAILED DESCRIPTION:
The goals of the PBM program:

* Improving patient care and optimizing blood management - quality assurance
* bleeding management based on latest scientific guidelines including:

  1. reduction of transfusion and better outcomes
  2. optimization of blood reserves
  3. introduction and acceptance of hospital protocols Previous research has identified gaps concerning implementation of PBM elements in CEE region calling for further research and training: anemia is not being managed appropriately, there are no protocols in place, patient journey is not clearly defined, it is not clear at which department should be anemia treated; availability of POC devices varies largely among countries; local protocols for management of severe bleeding are also missing in many hospitals.

Investigators plan to collect PBM implementation indicators in hospitals before PBM training at a given start point as baseline (first self audit) and re-evaluate achievements after 6 months after training (second self audit).

Investigators plan to define 2x1 week "snapshot" period for detailed analysis of perioperative approach at patient level (1 week at the beginning of the study and 1 week after 6 month).

Investigators assume that properly conducted self-audits followed by PBM training, optimizing local protocols and patient journeys, a reduction in the use of perioperative blood products may be achieved, which, in addition to the currently experienced decrease in the desire to donate blood, may lead to a more rational blood product management and better patient outcomes.

PBM Implementation indicators for hospitals (data to be collected):

* PBM administration & training data - are there PBM managers/local protocols available? was there any PBM training of staff performed?
* Pilar I.: data about diagnosis and management of anemia; patient pathways; medications used to treat anemia
* Pilar II.: blood saving techniques; usage of blood products (transfusion) and/or factor concentrates; iatrogenic blood loss - lab test tubes size
* Pilar III.: RBC tranfusion triggers;

Patient level data:

* age, gender, type of surgical intervention
* data about anemia management (performed or not by whom, when and what treatment was received if any
* data about existing anticoagulant therapy an management
* data about bleeding management (blood loss, transfusion requirements, factor concentrates (used quantities per routine medical intervention), POC tests evaluations if any, and standard laboratory test performed per routine medical approach before, during and after surgery
* data about postoperative outcomes

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years of age
* patients undergoing elective medium and high bleeding risk surgical intervention defined as moderate (<500 ml) and high (≥ 500 ml)
* patient consent

Exclusion Criteria:

* no patient consent
* patients under 18 years of age
* pregnant patients
* surgery with a low risk of bleeding
* the patient underwent emergency (non-elective) surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgerical interventions with medium or high bleeding risk during predefined two times one week periods - one week at basline and one week after 6 months
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Was the PBM training able to significantly reduce the use of blood products in the audited periods? | second self audit versus first self audit ( 6 months)
  Identification of local and country level PBM gaps during the first self audit followed by training and corrective measures, reidentification of remaining local and country level PBM gaps during the second self audit:
  1. Reduction of RBC, FFP and TC in Units
  2. PBM trained physichian in number

SECONDARY OUTCOMES:
Material assets for the PBM pillars | second self audit versus first self audit ( 6 months)
  1. increase in use of POC tests (number of tests)
  2. increase in use of factor concentrates (IU)
  3. local hemostasis management protocols (YES/NO)
Impact of PBM implementation on postoperative care | second self audit versus first self audit ( 6 months)
  Time spent in the intensive care unit in the postoperative period (ICU days)
Impact of PBM implementation on postoperative care | second self audit versus first self audit ( 9 months)
  Hospital length of stay (days)
PBM implementation impact on infection rates | second self audit versus first self audit ( 6 months)
  Postoperative infection rate
PBM implemetnation impact on mortality | second self audit versus first self audit ( 6 months)
  30 days mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meybohm P, Schmitt E, Choorapoikayil S, Hof L, Old O, Muller MM, Geisen C, Seifried E, Baumhove O, de Leeuw van Weenen S, Bayer A, Friederich P, Brautigam B, Friedrich J, Gruenewald M, Elke G, Molter GP, Narita D, Raadts A, Haas C, Schwendner K, Steinbicker AU, Jenke DJ, Thoma J, Weber V, Velten M, Wittmann M, Weigt H, Lange B, Herrmann E, Zacharowski K; German Patient Blood Management Network Collaborators. German Patient Blood Management Network: effectiveness and safety analysis in 1.2 million patients. Br J Anaesth. 2023 Sep;131(3):472-481. doi: 10.1016/j.bja.2023.05.006. Epub 2023 Jun 26. PMID 37380568
- [Background] Mitra B, Jorgensen M, Reade MC, Keegan A, Holley A, Farmer S, Harvey N, Winearls J, Parr M, French CJ; Clinical and Consumer Reference group for the update of Patient Blood Management Guidelines (Module 1: Critical Bleeding/Massive Transfusion). Patient blood management guideline for adults with critical bleeding. Med J Aust. 2024 Mar 4;220(4):211-216. doi: 10.5694/mja2.52212. Epub 2024 Jan 28. PMID 38282333
- [Background] Babik B, Fazakas J, Matusovits A, Gal J, Fulesdi B. [Perioperative Patient Blood Management: common risk, common tasks, common responsibility]. Orv Hetil. 2020 Sep;161(37):1545-1553. doi: 10.1556/650.2020.31918. Hungarian. PMID 32894734
- [Background] Olah Z, Fulesdi B, Gal J, Matusovits A, Babik B. [Principles of the perioperative Patient Blood Management]. Orv Hetil. 2020 Sep;161(37):1554-1568. doi: 10.1556/650.2020.31787. Hungarian. PMID 32894735
- [Background] Delaforce A, Duff J, Munday J, Hardy J. Preoperative Anemia and Iron Deficiency Screening, Evaluation and Management: Barrier Identification and Implementation Strategy Mapping. J Multidiscip Healthc. 2020 Dec 1;13:1759-1770. doi: 10.2147/JMDH.S282308. eCollection 2020. PMID 33293819
- [Background] Farmer SL, Towler SC, Leahy MF, Hofmann A. Drivers for change: Western Australia Patient Blood Management Program (WA PBMP), World Health Assembly (WHA) and Advisory Committee on Blood Safety and Availability (ACBSA). Best Pract Res Clin Anaesthesiol. 2013 Mar;27(1):43-58. doi: 10.1016/j.bpa.2012.12.007. PMID 23590915
- [Background] Hofmann A, Spahn DR, Holtorf AP; PBM Implementation Group. Making patient blood management the new norm(al) as experienced by implementors in diverse countries. BMC Health Serv Res. 2021 Jul 2;21(1):634. doi: 10.1186/s12913-021-06484-3. PMID 34215251
- [Background] Kietaibl S, Ahmed A, Afshari A, Albaladejo P, Aldecoa C, Barauskas G, De Robertis E, Faraoni D, Filipescu DC, Fries D, Godier A, Haas T, Jacob M, Lance MD, Llau JV, Meier J, Molnar Z, Mora L, Rahe-Meyer N, Samama CM, Scarlatescu E, Schlimp C, Wikkelso AJ, Zacharowski K. Management of severe peri-operative bleeding: Guidelines from the European Society of Anaesthesiology and Intensive Care: Second update 2022. Eur J Anaesthesiol. 2023 Apr 1;40(4):226-304. doi: 10.1097/EJA.0000000000001803. PMID 36855941
- [Background] Musallam KM, Tamim HM, Richards T, Spahn DR, Rosendaal FR, Habbal A, Khreiss M, Dahdaleh FS, Khavandi K, Sfeir PM, Soweid A, Hoballah JJ, Taher AT, Jamali FR. Preoperative anaemia and postoperative outcomes in non-cardiac surgery: a retrospective cohort study. Lancet. 2011 Oct 15;378(9800):1396-407. doi: 10.1016/S0140-6736(11)61381-0. Epub 2011 Oct 5. PMID 21982521
- [Background] Yan T, Lei S, Zhou B, Huang Y, Li X, Zhang J, Huang Q, Zhang L. Association between preoperative anemia and postoperative short-term outcomes in patients undergoing colorectal cancer surgery - a propensity score matched retrospective cohort study. BMC Anesthesiol. 2023 Sep 11;23(1):307. doi: 10.1186/s12871-023-02270-2. PMID 37697231
- [Background] Uden H, Buttner F, von Heymann C, Kramer M, Kaufner L, Vorderwulbecke G, Hardt S, Kruppa J, Balzer F, Spies C. Allogeneic Blood Transfusion and Risk of Postoperative Complications in Patients with Mild and Moderate Anemia of Any Cause? A Retrospective Cohort Study in Total Revision Hip Surgery. Transfus Med Hemother. 2023 Jul 12;51(1):12-21. doi: 10.1159/000530135. eCollection 2024 Feb. PMID 38314244
- See also: WHO PBM policy — https://www.who.int/publications/i/item/9789240035744
- See also: EU Publication office: practical PBM implementation guide for hospitals — https://op.europa.eu/en/publication-detail/-/publication/93e1bbbf-1a8b-11e7-808e-01aa75ed71a1/language-en
- See also: Information about PBM — https://patientbloodmanagement.org/learn/what-is-patient-blood-management/